CLINICAL TRIAL: NCT04895475
Title: Antibody Detection of Vaccine-Induced Secretory Effects
Acronym: ADVISE
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: ADVISE
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Covid19; Humoral Acquired Immunodeficiency; Coronavirus; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast milk: A small amount of breast milk (up to 10 mL) will be collected by the mother and frozen for future analysis. One breast milk sample per week is requested during the first eight weeks of study participation or until 3 months after the final vaccine dose (whichever is longer). Samples can be provided at an increased frequency (up to five times per week) in special circumstances such as a recent COVID infection or childbirth, or off schedule at the time of weaning, at the request of the PI.
  Blood: Finger-stick blood samples will be collected from study participants at baseline and then every two weeks for four consecutive samples or until 3 months after the final vaccine dose (whichever is longer) for serologic testing. Blood will be collected monthly from 3 through 6 months after final vaccination, and quarterly thereafter. Volumes of blood will be up to 0.5 mL at each collection, using small-sample Mitra devices from a finger stick.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lactating Mothers: Lactating mothers who plan to receive or have received the SARS-CoV-2 vaccine within 60 days.
  Interventions: Behavioral: SARS-CoV-2 vaccine

INTERVENTIONS:
Behavioral: SARS-CoV-2 vaccine — Baseline demographics, baseline breast milk samples, and blood collection will be obtained at the initial visit. Serial collections of breastmilk and blood as well as weekly self-administered monthly surveys will occur

SUMMARY:
The purpose of this research study is to conduct a prospective longitudinal surveillance research study, enrolling approximately 60 lactating mothers who receive the SARS-CoV-2 vaccine, and then following their clinical and laboratory parameters for up to 12 months. The overall goal is to investigate the characteristics of antibody formation in lactating women receiving SARS-CoV-2 vaccination, documenting the antibody isotypes, titers, duration, and transfer into milk over time.

DETAILED DESCRIPTION:
As the global and pandemic spread of the novel coronavirus (SARS-CoV-2, COVID-19) continues, many knowledge gaps remain regarding the epidemiology and transmission of infection, the immunological responses after viral exposure, and the immunological protection after vaccine administration. Cincinnati had its first confirmed case of COVID-19 on March 14, 2020, and despite extensive shelter-in-place and social distancing efforts, community spread has continued over the past 10 months with several distinct infection surges. As SARS-CoV-2 vaccines are becoming available in early 2021, it is important to understand the immunological effects of these vaccines and to contrast them to the effects of natural infection. Of particular interest are the immunological effects of SARS-CoV-2 vaccines for lactating women, and whether breast milk will include secretory antibodies against the virus that potentially confer protection to the breastfeeding infant. The investigators have a unique but time-limited opportunity to track the humoral immunological responses of SARS-CoV-2 vaccination among lactating women. The investigators designed Antibody Detection of Vaccine-Induced Secretory Effects (ADVISE) to collect and analyze serial breast milk samples for secretory antibody responses, along with periodic blood testing of the mothers and their breastfeeding children. In ADVISE, the investigators will document the prevalence and cumulative incidence of secretory antibody responses to SARS-CoV-2 vaccines, and gain insights into the protective immunological effects of elective vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18.0 years at the time of enrollment
* Currently lactating mothers
* Planning to receive the SARS-CoV-2 vaccine in the next 60 days, or vaccinated with the SARS-CoV-2 vaccine within the past 60 days
* Cell phone that can be used for text messaging or web-based viewing of surveys
* Willing and able to provide informed consent
* Ability to comply with all study related evaluations and follow-up

Exclusion Criteria:

* Any condition or illness that makes study participation ill-advised

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lactating mothers receiving the SARS-CoV-2 (COVID-19) vaccine.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
IgA antibodies against Spike protein | 12 months
  A 3-month cumulative prevalence of IgA antibodies against Spike protein after the completed administration of the SARS-CoV-2 vaccine.

SECONDARY OUTCOMES:
SARS-CoV-2 antibodies | 12 months
  The associations between maternal serum antibodies (onset, titer, duration) and breast milk antibodies against SARS-CoV-2, as well as comparisons of antibody responses after vaccine to natural infection.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Julie Ware, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ware J, McElhinney K, Latham T, Lane A, Dienger-Stambaugh K, Hildeman D, Spearman P, Ware RE. Sustained and Boosted Antibody Responses in Breast Milk After Maternal SARS-CoV-2 Vaccination. Breastfeed Med. 2023 Aug;18(8):612-620. doi: 10.1089/bfm.2023.0106. PMID 37615566